CLINICAL TRIAL: NCT05865912
Title: A Feasibility Study of Mindfulness Training Transcranial Direct Current Stimulation (tDCS) in Adults With Overweight and Obesity.
Acronym: MINDED
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: King's College London (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 3159550
Record Dates: First submitted 2023-04-11; First posted 2023-05-19 (Actual); Last update posted 2025-07-28 (Actual); Status verified 2023-04

CONDITIONS: Adults With Overweight and Obesity
Keywords: Mindfulness, Transcranial Direct Current Stimulation
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- [Mindfulness training + real tDCS] (Experimental)
  Interventions: Combination Product: Mindfulness training + real tDCS
- [Mindfulness training + sham tDCS] (Placebo Comparator)
  Interventions: Combination Product: Mindfulness training + sham tDCS
- [Waiting list control group]. (No Intervention)

INTERVENTIONS:
Combination Product: Mindfulness training + real tDCS — The MT is an established app-based programme delivered by Headspace®. During MT, participants complete guided meditation sessions which focus on mindful eating and on coping with cravings. Each MT session lasts 15 min. Participants in the MT+ real tDCS and MT+ sham tDCS groups will be given instructions to practice daily mindfulness for 3 weeks. During 10 of these sessions, MT and real/sham tDCS will be delivered concurrently.
  TDCS: During tDCS, a constant weak direct current is applied via electrodes (anode and cathode) placed on the scalp. In this study, the anode will be placed over the right dorsolateral prefrontal cortex (dlPFC) and the cathode will be placed over the left dlPFC. In the real tDCS condition, stimulation will be delivered at a constant current of 2 mA with a 10 second fade in/fade out for 20 minutes. In sham tDCS, the stimulator will deliver 60 seconds of active stimulation at the start ("ramping up") and end ("ramping down") of the 20 minute period.
  Arms: [Mindfulness training + real tDCS]
Combination Product: Mindfulness training + sham tDCS — Mindfulness training + sham tDCS
  Arms: [Mindfulness training + sham tDCS]

SUMMARY:
This study will investigate the feasibility of combining an app-based Mindfulness training (MT) with at-home administered transcranial direct current stimulation (tDCS) in adults with overweight or obesity and assess whether MT with tDCS may improve weight-related behaviours in this population. Specifically, the study will assess whether MT+ active tDCS, as opposed to MT+ sham tDCS or waiting list control, reduces high calorie food craving and consumption. Findings will inform the development of a future large-scale randomised controlled trial. The trial will be conducted in the UK.

DETAILED DESCRIPTION:
A randomised controlled feasibility trial with three parallel arms: [MT + real tDCS] vs [MT + sham tDCS] vs [Waiting list control group].

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 to 60 w
* Overweight or obese (BMI ≥25 kg/ m2) according to World Health Organisation (WHO) criteria.
* Use and understand English as a language for everyday conversation.
* Have access to a laptop or desktop computer with webcam and to able to attend baseline, post intervention and follow up assessments in the Institute of Psychiatry, Psychology and Neuroscience (KCL).

Exclusion Criteria:

* Insufficient written and spoken English
* All known contraindications to tDCS (Brunoni et al., 2012)
* Pregnancy; history of neurological disease and/or seizure
* Having any metallic implants in the head or body
* History of head or eye injury
* Significant health problems in the previous six months
* A lifetime diagnosis of substance dependence, psychosis, bipolar disorder, borderline personality disorder; any other primary psychiatric disorder requiring treatment in its own right
* Taking psychotropic medication
* Taking medication for weight loss Regular, current or past, mindfulness meditation or yoga practice (defined as > 20 minutes, twice or more per week during the past 2 months)
* Consuming more than 14 units of alcohol per week who are unwilling to reduce their alcohol intake for the duration of the treatment
* Current illicit drug use
* Learning difficulties that would preclude safe tDCS self-administration and/or completion of questionnaire measures and neurocognitive tasks (e.g.; working memory and inhibitory control)
* Current atypical anorexia nervosa or purging once a week or more.

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 52 (Actual)
Dates: Start 2023-10-17 (Actual); Primary Completion 2025-02-19 (Actual); Study Completion 2025-02-19 (Actual)

PRIMARY OUTCOMES:
The feasibility of combining an app-based Mindfulness training (MT) with at-home Administered transcranial direct current stimulation (tDCS) by assessing intervention adherence | post treatment assessment (assessed at week 3 post start of treatment)
  By assessing the tDCS session completed and the number of the MT sessions completed will be tracked through the app across the full 8 weeks
The feasibility of combining an app-based Mindfulness training (MT) with at-home Administered transcranial direct current stimulation (tDCS) by assessing intervention recruitment rate | post treatment assessment (assessed at week 3 post start of treatment)
  Recruitment rate/month over months will be assessed to demonstrate that recruitment targets for the main trial can be met within an adequate time-frame.
The feasibility of combining an app-based Mindfulness training (MT) with at-home Administered transcranial direct current stimulation (tDCS) by assessing intervention retention rates | post treatment assessment (assessed at week 3 post start of treatment) and at follow up (assessed at week 8 post start of treatment)
  determine retention rates from randomization through intervention completion
Participant views about treatment acceptability | post treatment assessment (assessed at week 3 post start of treatment)
  Treatment Acceptability Questionnaire: asking participants to indicate if MT with self-administered tDCS is an acceptable approach to treatment and whether they would recommend MT + tDCS to a friend if they were struggling with their weight.

SECONDARY OUTCOMES:
Change in high calorie food intake in the lab | Baseline assessment, post treatment assessment (assessed at week 3 post start of treatment) and at follow up up (assessed at week 8 post start of treatment)
  Taste Test: actual food consumption will be measured by means of a bogus "taste test". Consumption will be determined by weighing the food before and after the "taste test" and the difference in weight from pre- to post-assessment will be converted into calories and used as a measure of food intake.
Change in food cravings | Baseline assessment, post treatment assessment (assessed at week 3 post start of treatment) and at follow up up (assessed at week 8 post start of treatment)
  Food Cravings Questionnaire- Trait Version: it measures habitual experiences of food craving .
Change in weight loss using the bioelectrical impedance machine | Baseline assessment, post treatment assessment (assessed at week 3 post start of treatment) and at follow up up (assessed at week 8 post start of treatment)
  Body Mass Index will be calculated measuring body weight and height (kg/m2) using a bioelectrical impedance machine (InBody S10).
Change in emotion regulation using Emotion Regulation Questionnaire | Baseline assessment, post treatment assessment (assessed at week 3 post start of treatment) and at follow up up (assessed at week 8 post start of treatment)
  Emotion Regulation Questionnaire: A 10-item scale designed to measure respondents' tendency to regulate their emotions
Change in mood using the The Depression, Anxiety and Stress-Scale | Baseline assessment, post treatment assessment (assessed at week 3 post start of treatment) and at follow up up (assessed at week 8 post start of treatment)
  The Depression, Anxiety and Stress-Scale: is a 21-item self-report questionnaire which evaluates mood, anxiety and stress levels over the previous week.
Change in working memory | Baseline assessment, post treatment assessment (assessed at week 3 post start of treatment) and at follow up up (assessed at week 8 post start of treatment)
  Digital Span: the digit-span test for working memory is used to assess short-term memory. It has two subtests, the forward and backward tests.
Change in inhibitory control using the Go no Go Task | Baseline assessment, post treatment assessment (assessed at week 3 post start of treatment) and at follow up up (assessed at week 8 post start of treatment)
  Go no Go Task: this task measures response inhibition. In the go/no-go task, participants respond to certain stimuli ("go" stimuli) and make no response for others ("no-go" stimuli). The main dependent measure in go/no-go tasks is the commission error rate (making a "go" response on "no-go" trials); fewer errors signify better response inhibition.
Change mindful eating-related outcomes | Baseline assessment, post treatment assessment (assessed at week 3 post start of treatment) and at follow up up (assessed at week 8 post start of treatment)
  The Mindful Eating Questionnaire: is a 28-item questionnaire which will be used to assess awareness, distraction, disinhibition of eating and emotional and external eating. The
Change in food cravings using the Power of Food Scale | Baseline assessment, post treatment assessment (assessed at week 3 post start of treatment) and at follow up up (assessed at week 8 post start of treatment)
  Power of Food Scale: this assesses the psychological influence of the presence or Availability of food. It measures appetite for, rather than consumption of, palatable foods at three levels of food proximity (food available, food present, and food tasted)
Change in Body composition | Baseline assessment, post treatment assessment (assessed at week 3 post start of treatment) and at follow up up (assessed at week 8 post start of treatment)
  Body composition (primarily body fat percentage) will be assessed using a bioelectrical impedance machine (InBody S10).
Change in mood using Positive and Negative Affect Schedule | Baseline assessment, post treatment assessment (assessed at week 3 post start of treatment) and at follow up up (assessed at week 8 post start of treatment)
  Positive and Negative Affect Schedule: this consists of two 10-item self-report scale which measures positive and negative affect.
Change in inhibitory control using Barrett Impulsiveness Scale | Baseline assessment, post treatment assessment (assessed at week 3 post start of treatment) and at follow up up (assessed at week 8 post start of treatment)
  Barrett Impulsiveness Scale: this 30-item questionnaire during which participants are asked to reflect on a series of statements and indicate how frequently they apply to them.
Change in inhibitory control using Delayed Gratification Inventory | Baseline assessment, post treatment assessment (assessed at week 3 post start of treatment) and at follow up up (assessed at week 8 post start of treatment)
  Delayed Gratification Inventory: this questionnaire assesses participants' ability/tendency to delay gratification.
Change in mindfulness outcomes | Baseline assessment, post treatment assessment (assessed at week 3 post start of treatment) and at follow up up (assessed at week 8 post start of treatment)
  Mindful Awareness and Attention Scale: is a 15-item scale used to assess core characteristics of mindfulness
Eating Disorder Symptoms | Baseline assessment, post treatment assessment (assessed at week 3 post start of treatment) and at follow up up (assessed at week 8 post start of treatment)
  The Eating Disorder Examination Questionnaire (EDE-Q) will be used to assess eating disorders symptoms. The EDE-Q is a 36-item self-report quesitonnaire, and a higher global score indicates more severe eating disorder symptoms.

CONTACTS AND LOCATIONS:
Locations (1):
- CREW, London, Uk, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ageeli M, Flynn M, Lopes M, Ince B, Alves D, Westwood SJ, Campbell IC, Schmidt U. A feasibility study of the effects of concurrent transcranial direct current stimulation (tDCS) on mindfulness training in adults living with overweight or obesity: the MINDED trial protocol. Pilot Feasibility Stud. 2026 Jan 6;12(1):19. doi: 10.1186/s40814-025-01748-9. PMID 41495839